CLINICAL TRIAL: NCT06714799
Title: Analysis of Videodermatoscopic Parameters of Ocular, Periocular, Conjunctival and Palpebral Neoformations
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DER-OCCHI-19-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Ocular Surface Disease
Keywords: videodermatoscopia; occhi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ANALYSIS OF VIDEODERMATOSCOPIC PARAMETERS OF OCULAR, PERIOCULAR, CONJUNCTIVAL AND PALPEBRAL NEOFORMATIONS

DETAILED DESCRIPTION:
The analysis of videodermatoscopic parameters of ocular, periocular, conjunctival and eyelid neoformations refers to the use of advanced technology that allows us to examine in detail the lesions or neoformations that appear in and around the eye areas. Through videodermatoscopy, we can evaluate characteristics such as size, shape, color and internal structure of these neoformations, to distinguish benign ones from those that may require further diagnostic investigations or treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been diagnosed with one of the following conditions in the ocular and periocular region: common melanocytic nevus, melanosis, seborrheic keratosis, viral wart, angioma and angiokeratoma, apocrine hydrocystoma, xanthelasma, steatocystoma, actinic keratosis, basal cell carcinoma, squamous cell carcinoma, melanoma.

Exclusion Criteria:

* Patients who presented with one of the following conditions were excluded from the study: concomitant inflammatory processes, including blepharitis, chalazion, pterygium, pinguecula), coexistence of multiple, periocular or ocular lesions, diagnosis of syndromic diseases related to a major risk for cutaneous neoformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presented to the Videodermatoscopy Outpatient Clinic of the O.U. Dermatology of the S. Orsola-Malpighi General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
features that could indicate their benign or malignant nature | from enrollment to the end of 2026
  clinical and dermoscopic characteristics of periocular and ocular lesions

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Vaccari, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy